CLINICAL TRIAL: NCT05036447
Title: Recovery After Moderate-Heavy Resistance Exercise in Myotonic Dystrophy Type 1-patients
Brief Title: Myotonic Dystrophy Type 1 and Resistance Exercise
Acronym: STYRK DM1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Oslo University Hospital (Other); University of Southern Denmark (Other); University of Copenhagen (Other); Maastricht University (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Truls Raastad, Professor, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: STYRK DM1
Record Dates: First submitted 2021-05-10; First posted 2021-09-05 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Myotonic Dystrophy 1
Keywords: Resistance exercise; Recovery; Muscle protein synthesis; Muscle protein breakdown; Muscle function
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Intervention Model Description: Participants in both groups (patients and control) perform unilateral leg resistance exercise, contralateral leg serves as control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DM1-Ex (Experimental): Moderate-heavy resistance exercise of one leg in DM1-patients
  Interventions: Other: Moderate-Heavy Resistance Exercise
- DM1-Rest (No Intervention): Control leg (i.e. no exercise) in DM1-patients
- Ctrl-Ex (Experimental): Moderate-heavy resistance exercise of one leg in healthy participants
  Interventions: Other: Moderate-Heavy Resistance Exercise
- Ctrl-Rest (No Intervention): Control leg (i.e. no exercise) in healthy participants

INTERVENTIONS:
Other: Moderate-Heavy Resistance Exercise — Leg press: 3 x 8 repetitions at 75% of 1 repetition maximum, 3 minutes rest between sets.
  Knee extension: 3 x 6 repetitions at 85% of 1 repetition maximum, 3 minutes rest between sets.
  Arms: Ctrl-Ex; DM1-Ex

SUMMARY:
The purpose of this study is to investigate the response after one bout of moderate-heavy resistance exercise in patients suffering from Myotonic Dystrophy type 1. There is still doubt about if these patients could benefit from resistance exercise, or if this mode of exercise is detrimental to their mobility and health. We aim to monitor the subjects during the recovery phase and investigate recovery in several ways.

DETAILED DESCRIPTION:
Myotonic dystrophy type 1 (DM1) is an autosomal, dominantly inherited, muscular disease and the most common muscular dystrophy amongst adults. The disease is characterized by progressive myopathy and myotonia, first evident in the distal parts of the body: calves and forearms, further progressing towards proximal parts. A recent review by Voet and co-workers (2013) concludes that exercise is safe for DM1-patients, and based on our current knowledge, DM1-patients should be able to gain positive adaptations from exercise. However, the physiological outcomes of an exercise stimulus are not well studied in this population and because of alterations in important Ca2+ handling systems the recovery processes might be significantly different from healthy muscles.

The aim of this study is to investigate the acute responses to moderate-heavy resistance exercise in DM1-patients. We aim to establish a timeline for recovery of muscle strength, measured as maximal voluntary contraction. In line with this, we want to investigate if any muscular damage has occurred with both direct and indirect measures, and possible mechanisms leading to muscle damage, i.e. impaired Ca2+ handling.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Myotonic Dystrophy type 1-diagnosis

Exclusion Criteria:

* Non-ambulatory
* Injuries to muscle-skeletal-system that prevents resistance exercise
* Severe affection of the cardiovascular system
* Cognitive affection
* Lives more than one hour from test site

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in muscle strength | Baseline, and 5 minutes, 3 hours, 24 hours, 48 hours, and 71 hours after exercise
  Recovery of knee extension torque

SECONDARY OUTCOMES:
Muscle protein synthesis rate | Baseline and 27 hours after final session of resistance exercise
  Rate of muscle protein synthesis in m. vastus lateralis between baseline and 27 hours after final session of resistance exercise
Muscle protein breakdown rate | Baseline and 27 hours after final session of resistance exercise
  Rate of muscle protein breakdown in m. vastus lateralis between baseline and 27 hours after final session of resistance exercise

OTHER OUTCOMES:
Change in muscle damage | Baseline and 27 hours after final session of resistance exercise
  Myofibrillar disruption and necrosis observed in muscle tissue samples from m. vastus lateralis with electron microscopy
Change in muscle regeneration | Baseline and 27 hours after final session of resistance exercise
  Appearance of macrophages, satellite cell localization, and disruption of membrane in single muscle fibers and cross-sections using confocal microscopy
Change in calcium cycling | Baseline and 27 hours after final session of resistance exercise
  Calcium cycling in muscle tissue samples from m. vastus lateralis
Change in contractile function | Baseline and 27 hours after final session of resistance exercise
  Assessment of contractile function in single muscle fibers from m. vastus lateralis
Change in calcium-related protein abundances | Baseline and 27 hours after final session of resistance exercise
  Levels of protein and phosphorylation status using Western blotting
Muscle fiber type | Baseline
  Fiber type composition in samples from m. vastus lateralis
Muscle fiber type | 27 hours after final session of resistance exercise
  Fiber type composition in samples from m. vastus lateralis
Change in heat shock proteins | Baseline and 27 hours after final session of resistance exercise
  Localization and expression of heat shock proteins using Western blotting and Immunohistochemistry
Change in anabolic signaling | Baseline and 27 hours after final session of resistance exercise
  Expression and phosphorylation status of central mediators in anabolic signaling pathways using Western blotting
Change in autophagy | Baseline and 27 hours after final session of resistance exercise
  Expression and phosphorylation status of central mediators in pathways regulating muscle protein breakdown using Western blotting
Change in biomarkers of muscle damage | Baseline, and 3 hours, 24 hours, 48 hours, 71 hours, and 96 hours after exercise
  Levels of serum Creatine kinase, Myoglobin, and Troponin I
Change in biomarker of muscle damage | Baseline, and 20 hours, 44 hours, 68 hours, and 92 hours after exercise
  Level of titin-N fragment in urine
Change in Fatigue | Baseline, and 1 hour after exercise
  Electrical stimulation of m. vastus lateralis and m. vastus medialis at 10, 20, 50, and 80 Hz
Change in muscle stiffness | Baseline, and 50 minutes after exercise
  Muscle stiffness measured with shear wave elastography in static and dynamic conditions
Change in muscle soreness | Baseline, and 3 hours, 24 hours, 48 hours, and 71 hours after exercise
  Subjective rating of muscle soreness using a visual analogue scale (0-10)
Change in muscle swelling | Baseline, and 3 hours, 24 hours, 48 hours, and 71 hours after exercise
  Thickness of m. vastus lateralis using ultrasound B-mode

CONTACTS AND LOCATIONS:
Overall Officials: Truls Raastad, PhD, Principal Investigator — Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No